CLINICAL TRIAL: NCT00506896
Title: Monoarticular Corticosteroid Injection Versus Systemic Administration in the Treatment of Rheumatoid Arthritis Patients: A Randomized Double-Blind Controlled Study
Brief Title: Monoarticular Corticosteroid Injection Versus Systemic Administration in the Treatment of Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0599/04
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2007-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; glucocorticoid; intraarticular injection; arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Injections, Intra-Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: intraarticular injection

INTERVENTIONS:
Drug: intraarticular injection — Triamcinolone hexacetonide 60mg(3ml)by intraarticular injection Triamcinolone acetonide 60mg (3ml)by intramuscular administration
  Other Names: Triancil®; Theracort®

SUMMARY:
The purpose of this study is to compare the efficacy and safety of intra-articular glucocorticoid injection to its systemic use for treatment of knee synovitis in patients with Rheumatoid Arthritis

DETAILED DESCRIPTION:
A randomized double-blind controlled study was conducted including 60 patients with RA. Patients were randomized to receive either a single intra-articular knee injection with triamcinolone hexacetonide 60 mg and xylocaine chloride 2% (1 mL) associated to a single intramuscular injection of 1 mL of xylocaine chloride 2% (IAI group) or 1 mL of xylocaine chloride 2% by intra-articular injection and a intramuscular injection of triamcinolone acetonide 60 mg and xylocaine chloride 2% (1 mL) (IM group). Evaluations were performed at baseline and 1, 4, 8 and 12 weeks post-intervention. The following instruments were used: the ACR 20%, 50 and 70% improvement criteria; VAS for knee morning stiffness, pain and edema; knee circumference and goniometry; Likert's scale of improvement (IVAS); daily use of oral glucocorticoid and NSAIDs, blood pressure and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid Arthritis diagnosed for more than 6 months
* 18 and 65 years
* Functional class II or III according to the ACR criteria
* VAS for knee pain higher than 5
* Use of stable doses of oral corticosteroid for the last 30 days
* Use of stable doses of DMARDs for the last 3 months
* Active synovitis at least in one knee for at least the 30 days

Exclusion Criteria:

* Non-controlled diabetes mellitus or hypertension
* Bacterial infection of any site
* Blood coagulation disorders
* Skin lesion on the affected knee
* History of previous surgical procedure in the knee
* Use of intra-muscular glucocorticoid in the last 30 days
* Intra-articular injection in the last 3 months
* Knee injection in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-07; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
VAS for knee pain | 12 weeks post intervention

SECONDARY OUTCOMES:
side and adverse effects, safety | 12 weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Monique S Konai, MD, Principal Investigator — Federal University of São Paulo; Rita V Furtado, MD, PhD, Study Director — Federal University of São Paulo; Marla F Santos, MD, Principal Investigator — Federal University of São Paulo; Jamil Natour, MD, PhD, Study Chair — Federal University of São Paulo
Locations (1):
- Rheumatology Division, Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Gray RG, Gottlieb NL. Intra-articular corticosteroids. An updated assessment. Clin Orthop Relat Res. 1983 Jul-Aug;(177):235-63. PMID 6345042
- [Background] Verstappen SM, Jacobs JW, Bijlsma JW; Utrecht Rheumatoid Arthritis Cohort Study Group. The Utrecht experience with different treatment strategies in early rheumatoid arthritis. Clin Exp Rheumatol. 2003 Sep-Oct;21(5 Suppl 31):S165-8. PMID 14969070
- [Background] See Y. Intra-synovial corticosteroid injections in juvenile chronic arthritis--a review. Ann Acad Med Singap. 1998 Jan;27(1):105-11. PMID 9588284
- [Background] Caldwell JR. Intra-articular corticosteroids. Guide to selection and indications for use. Drugs. 1996 Oct;52(4):507-14. doi: 10.2165/00003495-199652040-00004. PMID 8891463
- [Background] Bird HA, Ring EF, Daniel R, Bacon PA. Comparison of intra-articular methotrexate with intra-articular triamcinolone hexacetonide by thermography. Curr Med Res Opin. 1977;5(2):141-6. doi: 10.1185/03007997709110154. PMID 340129
- [Background] Marchesoni A, Sinigaglia L, Ranza R, Varenna M, Battafarano N, Tosi S. Rifamycin SV versus triamcinolone in local treatment of rheumatoid synovitis. Scand J Rheumatol. 1993;22(4):194-8. doi: 10.3109/03009749309099270. PMID 8356413
- [Background] Stein A, Yassouridis A, Szopko C, Helmke K, Stein C. Intraarticular morphine versus dexamethasone in chronic arthritis. Pain. 1999 Dec;83(3):525-532. doi: 10.1016/S0304-3959(99)00156-6. PMID 10568861
- [Background] Schatteman L, Gyselbrecht L, De Clercq L, Mielants H. Treatment of refractory inflammatory monoarthritis in ankylosing spondylitis by intraarticular injection of infliximab. J Rheumatol. 2006 Jan;33(1):82-5. Epub 2005 Nov 15. PMID 16292792
- [Background] Bliddal H, Terslev L, Qvistgaard E, Konig M, Holm CC, Rogind H, Boesen M, Danneskiold-Samsoe B, Torp-Pedersen S. A randomized, controlled study of a single intra-articular injection of etanercept or glucocorticosteroids in patients with rheumatoid arthritis. Scand J Rheumatol. 2006 Sep-Oct;35(5):341-5. doi: 10.1080/03009740600844530. PMID 17062431
- [Background] Blyth T, Stirling A, Coote J, Land D, Hunter JA. Injection of the rheumatoid knee: does intra-articular methotrexate or rifampicin add to the benefits of triamcinolone hexacetonide? Br J Rheumatol. 1998 Jul;37(7):770-2. doi: 10.1093/rheumatology/37.7.770. PMID 9714355
- [Background] Hollander JL. Intra-synovial corticosteroid therapy in rheumatoid arthritis. MD Med J 1970;19:62-66.
- [Background] MCCARTY DJ Jr, FAIRES JS. A comparison of the duration of local anti-inflammatory effect of several adrenocorticosteroid esters--a bioassay technique. Curr Ther Res Clin Exp. 1963 May;5:284-90. No abstract available. PMID 13932060
- [Background] Derendorf H, Mollmann H, Gruner A, Haack D, Gyselby G. Pharmacokinetics and pharmacodynamics of glucocorticoid suspensions after intra-articular administration. Clin Pharmacol Ther. 1986 Mar;39(3):313-7. doi: 10.1038/clpt.1986.45. PMID 3948470
- [Background] Bain LS, Balch HW, Wetherly JM, Yeadon A. Intraarticular triamcinolone hexacetonide: double-blind comparison with methylprednisolone. Br J Clin Pract. 1972 Dec;26(12):559-61. No abstract available. PMID 4567862
- [Background] Bird HA, Ring EF, Bacon PA. A thermographic and clinical comparison of three intra-articular steroid preparations in rheumatoid arthritis. Ann Rheum Dis. 1979 Feb;38(1):36-9. doi: 10.1136/ard.38.1.36. PMID 373651
- [Background] Jalava S, Saario R. Treatment of finger joints with local steroids. A double-blind study. Scand J Rheumatol. 1983;12(1):12-4. doi: 10.3109/03009748309101996. PMID 6836233
- [Background] Blyth T, Hunter JA, Stirling A. Pain relief in the rheumatoid knee after steroid injection. A single-blind comparison of hydrocortisone succinate, and triamcinolone acetonide or hexacetonide. Br J Rheumatol. 1994 May;33(5):461-3. doi: 10.1093/rheumatology/33.5.461. PMID 8173851
- [Background] Zulian F, Martini G, Gobber D, Agosto C, Gigante C, Zacchello F. Comparison of intra-articular triamcinolone hexacetonide and triamcinolone acetonide in oligoarticular juvenile idiopathic arthritis. Rheumatology (Oxford). 2003 Oct;42(10):1254-9. doi: 10.1093/rheumatology/keg358. Epub 2003 Jun 16. PMID 12810938
- [Background] McCarty DJ. Treatment of rheumatoid joint inflammation with triamcinolone hexacetonide. Arthritis Rheum. 1972 Mar-Apr;15(2):157-73. doi: 10.1002/art.1780150205. No abstract available. PMID 5027603
- [Background] HOLLANDER JL, BROWN EM Jr, JESSAR RA, BROWN CY. Hydrocortisone and cortisone injected into arthritic joints; comparative effects of and use of hydrocortisone as a local antiarthritic agent. J Am Med Assoc. 1951 Dec 22;147(17):1629-35. doi: 10.1001/jama.1951.03670340019005. No abstract available. PMID 14880415
- [Background] Arnett FC, Edworthy SM, Bloch DA, McShane DJ, Fries JF, Cooper NS, Healey LA, Kaplan SR, Liang MH, Luthra HS, et al. The American Rheumatism Association 1987 revised criteria for the classification of rheumatoid arthritis. Arthritis Rheum. 1988 Mar;31(3):315-24. doi: 10.1002/art.1780310302. PMID 3358796
- [Background] Hochberg MC, Chang RW, Dwosh I, Lindsey S, Pincus T, Wolfe F. The American College of Rheumatology 1991 revised criteria for the classification of global functional status in rheumatoid arthritis. Arthritis Rheum. 1992 May;35(5):498-502. doi: 10.1002/art.1780350502. PMID 1575785
- [Background] Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, Katz LM, Lightfoot R Jr, Paulus H, Strand V, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995 Jun;38(6):727-35. doi: 10.1002/art.1780380602. PMID 7779114
- [Background] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777
- [Background] Lequesne MG. The algofunctional indices for hip and knee osteoarthritis. J Rheumatol. 1997 Apr;24(4):779-81. PMID 9101517
- [Background] McCarty DJ, Harman JG, Grassanovich JL, Qian C. Treatment of rheumatoid joint inflammation with intrasynovial triamcinolone hexacetonide. J Rheumatol. 1995 Sep;22(9):1631-5. PMID 8523335
- [Background] Srinivasan A, Amos M, Webley M. The effects of joint washout and steroid injection compared with either joint washout or steroid injection alone in rheumatoid knee effusion. Br J Rheumatol. 1995 Aug;34(8):771-3. doi: 10.1093/rheumatology/34.8.771. PMID 7551664
- [Background] Armstrong RD, English J, Gibson T, Chakraborty J, Marks V. Serum methylprednisolone levels following intra-articular injection of methylprednisolone acetate. Ann Rheum Dis. 1981 Dec;40(6):571-4. doi: 10.1136/ard.40.6.571. PMID 7332377
- [Background] Steer JH, Ma DT, Dusci L, Garas G, Pedersen KE, Joyce DA. Altered leucocyte trafficking and suppressed tumour necrosis factor alpha release from peripheral blood monocytes after intra-articular glucocorticoid treatment. Ann Rheum Dis. 1998 Dec;57(12):732-7. doi: 10.1136/ard.57.12.732. PMID 10070273
- [Background] Weitoft T, Ronnblom L. Randomised controlled study of postinjection immobilisation after intra-articular glucocorticoid treatment for wrist synovitis. Ann Rheum Dis. 2003 Oct;62(10):1013-5. doi: 10.1136/ard.62.10.1013. PMID 12972485
- [Background] Proudman SM, Conaghan PG, Richardson C, Griffiths B, Green MJ, McGonagle D, Wakefield RJ, Reece RJ, Miles S, Adebajo A, Gough A, Helliwell P, Martin M, Huston G, Pease C, Veale DJ, Isaacs J, van der Heijde DM, Emery P. Treatment of poor-prognosis early rheumatoid arthritis. A randomized study of treatment with methotrexate, cyclosporin A, and intraarticular corticosteroids compared with sulfasalazine alone. Arthritis Rheum. 2000 Aug;43(8):1809-19. doi: 10.1002/1529-0131(200008)43:83.0.CO;2-D. PMID 10943871
- [Background] Hetland ML, Stengaard-Pedersen K, Junker P, Lottenburger T, Ellingsen T, Andersen LS, Hansen I, Skjodt H, Pedersen JK, Lauridsen UB, Svendsen A, Tarp U, Podenphant J, Hansen G, Lindegaard H, de Carvalho A, Ostergaard M, Horslev-Petersen K; CIMESTRA Study Group. Combination treatment with methotrexate, cyclosporine, and intraarticular betamethasone compared with methotrexate and intraarticular betamethasone in early active rheumatoid arthritis: an investigator-initiated, multicenter, randomized, double-blind, parallel-group, placebo-controlled study. Arthritis Rheum. 2006 May;54(5):1401-9. doi: 10.1002/art.21796. PMID 16645967
- [Background] American College of Rheumatology Subcommittee on Rheumatoid Arthritis Guidelines. Guidelines for the management of rheumatoid arthritis: 2002 Update. Arthritis Rheum. 2002 Feb;46(2):328-46. doi: 10.1002/art.10148. No abstract available. PMID 11840435
- [Background] Intra-articular radioactive yttrium and triamcinolone hexacetonide: an inconclusive trial. Arthritis and Rheumatism Council Multicentre Radiosynoviorthesis Trial Group. Ann Rheum Dis. 1984 Aug;43(4):620-3. doi: 10.1136/ard.43.4.620. PMID 6383234
- [Background] Silverman E, Spiegel L, Hawkins D, Petty R, Goldsmith D, Schanberg L, Duffy C, Howard P, Strand V. Long-term open-label preliminary study of the safety and efficacy of leflunomide in patients with polyarticular-course juvenile rheumatoid arthritis. Arthritis Rheum. 2005 Feb;52(2):554-62. doi: 10.1002/art.20861. PMID 15693001
- [Background] Neidel J, Boehnke M, Kuster RM. The efficacy and safety of intraarticular corticosteroid therapy for coxitis in juvenile rheumatoid arthritis. Arthritis Rheum. 2002 Jun;46(6):1620-8. doi: 10.1002/art.10313. PMID 12115194
- [Background] Schumacher HR, Chen LX. Injectable corticosteroids in treatment of arthritis of the knee. Am J Med. 2005 Nov;118(11):1208-14. doi: 10.1016/j.amjmed.2005.05.003. PMID 16271901
- [Background] Ostergaard M, Stoltenberg M, Gideon P, Sorensen K, Henriksen O, Lorenzen I. Changes in synovial membrane and joint effusion volumes after intraarticular methylprednisolone. Quantitative assessment of inflammatory and destructive changes in arthritis by MRI. J Rheumatol. 1996 Jul;23(7):1151-61. PMID 8823685
- [Background] Weitoft T, Larsson A, Saxne T, Ronnblom L. Changes of cartilage and bone markers after intra-articular glucocorticoid treatment with and without postinjection rest in patients with rheumatoid arthritis. Ann Rheum Dis. 2005 Dec;64(12):1750-3. doi: 10.1136/ard.2004.035022. Epub 2005 Apr 20. PMID 15843449
- [Background] Huppertz HI, Pfuller H. Transient suppression of endogenous cortisol production after intraarticular steroid therapy for chronic arthritis in children. J Rheumatol. 1997 Sep;24(9):1833-7. PMID 9292813
- [Background] Kirwan JR. The effect of glucocorticoids on joint destruction in rheumatoid arthritis. The Arthritis and Rheumatism Council Low-Dose Glucocorticoid Study Group. N Engl J Med. 1995 Jul 20;333(3):142-6. doi: 10.1056/NEJM199507203330302. PMID 7791815
- [Background] Sholter DE, Armstrong PW. Adverse effects of corticosteroids on the cardiovascular system. Can J Cardiol. 2000 Apr;16(4):505-11. PMID 10787466
- [Background] Reid IR. Glucocorticoid-induced osteoporosis. Baillieres Best Pract Res Clin Endocrinol Metab. 2000 Jun;14(2):279-98. doi: 10.1053/beem.2000.0074. PMID 11035907
- [Background] Furtado RN, Oliveira LM, Natour J. Polyarticular corticosteroid injection versus systemic administration in treatment of rheumatoid arthritis patients: a randomized controlled study. J Rheumatol. 2005 Sep;32(9):1691-8. PMID 16142862
- [Background] Rausch-Stroomann JG, Petry R, Brandt T, Thomas E. [Comparative study on intramuscular and intraarticular administration of the depot steroid Triamcinolone acetonide]. Arzneimittelforschung. 1971 Jun;21(6):836-40. No abstract available. German. PMID 5109272
- [Background] Adebajo AO, Nash P, Hazleman BL. A prospective double blind dummy placebo controlled study comparing triamcinolone hexacetonide injection with oral diclofenac 50 mg TDS in patients with rotator cuff tendinitis. J Rheumatol. 1990 Sep;17(9):1207-10. PMID 2290163
- See also: Federal University of Sao Paulo — http://www.unifesp.br